CLINICAL TRIAL: NCT05115877
Title: Evaluation of Outcomes From Treatment of Benign or Malignant Gastrointestinal Diseases
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 031.HPB.2020.R
Record Dates: First submitted 2020-11-18; First posted 2021-11-10 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-04

CONDITIONS: Gastrointestinal Disease
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be a retrospective, registry study collecting data of patients who were diagnosed with benign or malignant gastrointestinal diseases. Data will be collected from patient's chart retrospectively once the patients have completed proper treatment follow up with physicians' practice.

DETAILED DESCRIPTION:
It is reported in the literature that the treatment of any gastrointestinal disease process, whether benign or malignant, continues to be a huge challenge. For example, patients with gastrointestinal cancer continue to be diagnosed at an advanced stage with medical and surgical options that are improving in terms of outcome measurements but with much more room for improvement. The goal is to continue to review our treatment outcomes to further improve overall survival, overall symptom control, mortality and morbidity.

The main aim of this study is to evaluate and compare the outcomes from our treatment of benign or malignant gastrointestinal diseases through medical chart review.

There is a need to understand and improve the current diagnosis and treatment algorithm for gastrointestinal pathologies. Continued evaluation and study is imperative to ensure that national guidelines are improving to enhance patient cure and/or recovery.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed and treated for gastrointestinal diseases, benign or malignant from 2005 to 2030.
* Age ≥18 years

Exclusion Criteria:

* Patients that are not diagnosed with or treated for gastrointestinal diseases
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with benign or malignant gastrointestinal diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2024-05-17 (Estimated); Study Completion 2024-05-17 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Jan 2005 - Jan 2030
  from day of diagnosis or procedure to death date
Overall symptom | Jan 2005 - Jan 2030
  Difficulty swallowing, Heartburn, Regurgitation, Chest pain, Weight Loss, Quality of life
Mortality | Jan 2005 - Jan 2030
  death or life
Morbidity | Jan 2005 - Jan 2030
  yes or no to individual disease

CONTACTS AND LOCATIONS:
Overall Officials: Dhiresh R Jeyarajah, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Richardson Medical Center, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No